CLINICAL TRIAL: NCT02800707
Title: Sucralose, Stevia, Gut Microbiome and Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 1605M88288
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — trichlorosucrose; stevioside

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sucralose (Active Comparator): Participants will be asked to consume 180 mg/day of sucralose (in the form of capsules which is equivalent to three 12-oz cans of diet soda) for 14 days. According to the FDA, a 150 lb. person may consume up to 340 mg/day of sucralose (or 5.5 12-oz cans of sucralose-sweetened diet soda).
  Interventions: Other: Sucralose
- Stevia (Active Comparator): Participants will be asked to consume 180 mg/day of stevia (in the form of capsules which is equivalent to three 12-oz cans of diet soda) for 14 days. According to the FDA, a 150 lb. person may consume up to 800 mg/day of stevia (or about 12 cans of stevia-sweetened diet soda).
  Interventions: Other: Stevia

INTERVENTIONS:
Other: Sucralose — Sweetner
  Arms: Sucralose
Other: Stevia — Sweetner
  Arms: Stevia

SUMMARY:
This study will determine the influence of two non-caloric sweeteners on glucose metabolism via the gut microbiome in adult men and women.

DETAILED DESCRIPTION:
This study will determine the influence of two non-caloric sweeteners on glucose metabolism via the gut microbiome in adult men and women aged 35-55 years.

ELIGIBILITY:
Inclusion Criteria: Generally health adult men and women aged 35-55 years old -

Exclusion Criteria:Adults will not be eligible who have chronic disease (cancer, CHD, diabetes, chronic kidney disease); pregnant or breast feeding; menopausal; has a history of bariatric surgery; taking prednisone/steroids, taking medication for PCOS, or take medications that influence blood glucose.

-

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-01-03 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
2-hour glucose | 14 days
  An oral glucose tolerance test will be administered before and after consuming assigned sweetener to determine change in 2-hour glucose

SECONDARY OUTCOMES:
Gut microbiome | 14 days
  Gut microbiota will be measured before and after consuming assigned sweetener to determine change in gut microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Lyn M Steffen, PhD, Principal Investigator — University of Minnesota
Locations (1):
- ECRC, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be made available.